CLINICAL TRIAL: NCT02794324
Title: Optimisation and Individualisation of Heart-Sparing Breast Radiotherapy Techniques (The HeartSpare Study)
Brief Title: The HeartSpare Study (Stage I)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCR3593
Record Dates: First submitted 2011-10-28; First posted 2016-06-09 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Voluntary deep-inspiratory breath hold (Experimental): Stage 1A: Voluntary deep-inspiratory breath hold (v_DIBH) vs Active-breathing-controlled deep-inspiratory breathhold (ABC_DIBH)
  Interventions: Procedure: Voluntary deep-inspiratory breath hold
- Active-breathing-controlled deep-inspiratory breathhold (Active Comparator): Stage 1A: Voluntary deep-inspiratory breath hold (v_DIBH) vs Active-breathing-controlled deep-inspiratory breathhold (ABC_DIBH)
  Interventions: Procedure: Active-breathing-controlled deep-inspiratory breathhold; Device: Active-breathing-controlled deep-inspiratory breathhold
- Prone treatment (Active Comparator): Stage 1B: Optimised supine DIBH vs prone position
  Interventions: Procedure: Prone treatment

INTERVENTIONS:
Procedure: Voluntary deep-inspiratory breath hold — Patients undergoing scanning in v_DIBH will be positioned supine with arms extended on a MedTec breast board. They will be monitored visually on screen and will be given a buzzer to press when they have taken a breath. CT images will be obtained during DIBH. If the patient needs to release their breath, they will be asked to press the buzzer a second time. Patients will be closely monitored by radiographers via CCTV.
  Arms: Voluntary deep-inspiratory breath hold
Procedure: Active-breathing-controlled deep-inspiratory breathhold — Patients undergoing scanning in ABC_DIBH will be positioned supine with arms extended on a MedTec breast board to which an activated-breathing control device (Elekta, Crawley, UK) has been attached. They will breathe through the device. During ABC_DIBH, CT images will be obtained.
  Arms: Active-breathing-controlled deep-inspiratory breathhold
Procedure: Prone treatment — Patients undergoing scanning in a prone position will lie on a customised prone treatment platform. CT images will be acquired under free-breathing conditions.
  Arms: Prone treatment
Device: Active-breathing-controlled deep-inspiratory breathhold — The ABC unit allows for temporary and reproducible immobilization of internal thoracic structures by monitoring the patient's breathing cycle and implementing a breath hold at a predefined lung volume level. The device consists of a mouthpiece connected to a pneumotachometer via a bidirectional valve and tubing. The air flow across the pneumotachometer is integrated and displayed on a computer monitor. The computer also controls a scissor valve which, when enabled, restricts air flow through the system, enabling the breath hold phase. The mouthpiece and air filter are patient specific, as is a nose clip that is used to ensure that patients are breathing through the device.
  Other Names: Active Breathing Coordinator (Elekta, Crawley, UK)
  Arms: Active-breathing-controlled deep-inspiratory breathhold

SUMMARY:
Radiotherapy (RT) has a major curative role in women with early breast cancer, and is recommended routinely after lumpectomy and selectively after mastectomy. It has contributed to a halving of breast cancer mortality in the UK over the last 2 decades despite ever-rising cancer incidence. RT in women with left-sided tumours often exposes the underlying heart to a damaging dose. The heart is very sensitive to RT, and there were 1-2 deaths from heart disease for every 100 breast cancer patients treated during the 1960s-70s. The situation has improved in recent years, but standard RT techniques still deliver significant radiation doses to heart tissue.

Two potentially simple techniques reduce heart dose. In one, women are taught to breathe in deeply and to hold their breath for about 20 seconds while RT is given. The downward movement of the diaphragm pulls the heart away from the RT beam. In the other technique, women lie on their fronts, instead of on their backs as they normally do for breast RT. In this position, the breast falls away from the rib cage and reduces exposure of the heart. Neither technique is routinely available to women receiving breast RT in the UK for reasons that this research aims to address. The investigators need to: 1) confirm that patient position can be reproduced with millimetre precision every day using these techniques, 2) minimise costs of equipment, time and personnel required to support such techniques, 3) select the most appropriate technique for different patients and 4) train staff in centres across the UK to deliver techniques safely and effectively. By addressing all of these issues, the study aims ultimately to make heart-sparing RT available to all UK women that might benefit from treatment, thereby significantly reducing the burden of heart disease in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Complete microscopic excision of early stage invasive ductal or lobular carcinoma (pT1-3b N0-1 M0) of the left breast following breast conservation surgery or mastectomy.
* Recommendation for whole breast (groups A and B) or chest wall (Group A only) radiotherapy (with or without tumour bed boost)
* Age ≥18
* Performance status ≤1
* Patients able to tolerate breath-hold

Exclusion Criteria:

* Requirement for nodal irradiation
* Patients with micro- or macro-scopic disease on sentinel node biopsy who have not undergone completion axillary node clearance
* Previous radiotherapy to any region above the diaphragm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Interfraction reproducibility of chest wall position (group A) | End of radiotherapy (3-4 weeks)
  The position of ipsilateral chest wall will be compared between the digitally reconstructed radiographs (derived from the planning CT) and the on-treatment electronic portal images and mean daily displacements calculated.
Difference in mean left anterior descending coronary artery (LAD) mean normal tissue dose (NTDmean) (group B) | End of radiotherapy (3-4 weeks)
  Using dose-volume histograms (DVHs) based on the planning scan and on-treatment CBCT imaging, mean LAD NTDmean will be compared for ABC_DIBH versus prone positioning.

SECONDARY OUTCOMES:
Difference in NTDmean for heart, LAD, ipsilateral and whole lungs (group A) | End of radiotherapy (3-4 weeks)
Comparison of standard deviation in mean LAD NTDmean over a treatment course (group B) | End of radiotherapy (3-4 weeks)
Comparison of individual patient heart NTDmean differences by anatomical factors (group B) | End of radiotherapy (3-4 weeks)
Difference in mean normal tissue doses (NTDmean) to heart, ipsilateral and whole lungs (group B) | End of radiotherapy (3-4 weeks)
Difference in volumes of chest wall receiving 20Gy (Groups A and B) | End of radiotherapy (3-4 weeks)
Interfraction reproducibility of chest wall position (groups A and B) | End of radiotherapy (3-4 weeks)
Interfraction reproducibility of tumour bed position (groups A and B) | End of radiotherapy (3-4 weeks)
Time and equipment costs (groups A and B) | End of study (2 years)
Patient and radiographer satisfaction with positioning technique (groups A and B) | Weekly questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kirby, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, United Kingdom